CLINICAL TRIAL: NCT06520150
Title: Evaluation of the Effectiveness of Two Methods of Regional Anesthesia During Subcutaneous Implantable Cardioverter-defibrillator (SICD) Implantation Procedure.
Brief Title: Evaluation of the Effectiveness of Two Methods of Regional Anesthesia During S-ICD Implantation Procedure.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Responsible Party: Principal Investigator, Marek Szamborski, Senior Assistant, MD, 4th Military Clinical Hospital with Polyclinic, Poland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 3_2024
Record Dates: First submitted 2024-07-08; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Chest Pain; Pain, Procedural; Pain, Postoperative; Analgesia; Regional Anesthesia Morbidity; Anesthesia, Local; ICD
Keywords: Superficial Serratus Anterior Plane Block (SSAP); Superficial Parasternal Intercostal Plane Block (SPIP); Pectoserratus Plane Blocks (PSP); Regional anaesthesia; Subcutaneous implantable defibrillator (S-ICD); thorax blockade; less invasive; implantation; pain treatment
MeSH Terms: conditions — Chest Pain; Pain, Procedural; Pain, Postoperative; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly divided into 2 groups - Group I will be patients administered PSP+SSAP anesthesia (consecutively 20+40ml of the mixture indicated above). Group II will be patients given SPIP+SSAP blockade (consecutively 20+40ml of the mixture indicated above). It was tentatively planned to conduct the study on a group of 32 patients (16 in each of the two groups).
Who Masked: Participant, Care Provider
Masking Description: Anesthesiologists administering anesthesia prior to surgery receive an envelope with a randomly indicated method of anesthesia based on simple randomization determines the type of regional blockade used during the procedure). The subject will not know which study group he or she has been classified into. The operator performing the procedure will not be informed of the type of anesthesia performed -[randomization by double-blinding]. The operator performing the procedure will not be informed about the type of block performed in order to objectivize the extent and quality of the subject's anesthesia, which he will evaluate after the procedure according to a scale of subjective operator comfort created (EOA scale).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (PSP+SSAP) (Active Comparator): Group I will include patients undergoing PSP(Pectoserratus plane block)+SSAP(Superficial serratus anterior plane block) (20+40ml) The solution is defined as a combination of 0.125% ropivacaine solution with 0.25% lidocaine solution in a total volume of 60ml of liquid administered.
  Interventions: Procedure: Regional anaesthetic combined fascial plane block; Drug: Ropivacaine 0.125% Injectable Solution +Lignocaine 0,25% Injectable Solution
- Group I (SPIP+SSAP) (Active Comparator): Group II will include patients undergoing SPIP(Superficial parastenal intercostal plane block)+SSAP(Superficial serratus anterior plane block) (20+40ml) The solution is defined as a combination of 0.125% ropivacaine solution with 0.25% lidocaine solution in a total volume of 60ml of liquid administered.
  Interventions: Procedure: Regional anaesthetic combined fascial plane block; Drug: Ropivacaine 0.125% Injectable Solution +Lignocaine 0,25% Injectable Solution

INTERVENTIONS:
Procedure: Regional anaesthetic combined fascial plane block — Prior to the procedure, the anaesthetists will receive an envelope from a person not related to the project (a hospital administrative staff member). This envelope will contain a randomly indicated method of anaesthesia based on simple randomisation. This will determine the type of regional block used during the procedure. It is important to note that the patient will not know which study group they have been classified in. Furthermore, the operator performing the procedure will not be informed of the type of anaesthesia performed. This is to ensure double-blinding. In order to ensure the highest standards of objectivity, the operator performing the procedure will not be informed about the type of block performed. This will allow us to assess the extent and quality of anaesthesia after the procedure, We will use a proprietary scale of subjective operator comfort scale.
  Other Names: PSP; SPIP; SSAP
Drug: Ropivacaine 0.125% Injectable Solution +Lignocaine 0,25% Injectable Solution — administration under ultrasound guidance of a mixture of 2 local anaesthetics in a fixed total volume

SUMMARY:
Our study consists of a combination of regional blockade ('local' anesthesia) of the anterior and lateral chest wall in the form of a thin needle prick and the supply of local anesthetic drugs to the area of the relevant chest wall structures to exclude all stimuli, including pain from the operative site. A short-acting analgesic and sedative drug will be administered intravenously throughout the procedure - in a dose that allows the required contact between the patient and the anesthetist. If necessary, the dose of the drug may be increased to maintain pain comfort throughout the procedure.

The anesthetic team will be with the patient throughout the procedure to ensure comfort and safety.

DETAILED DESCRIPTION:
The current study is a continuation of the 2021-2023 project, during which 16 patients were anesthetized using a combination of previously known regional (PSP +SSAP) blocks in the thoracic area for S-ICD implantation. PSP (pectoserratus plane) block, previously known in scientific nomenclature as (PECS II /DPP/ PNB II) is a block placed under the pectoralis minor muscle between the pectoralis anterior muscle or also under it in the area of the III/IV rib lateral to the midclavicular line. SSAP (superficial serratus anterior plane) block is formerly known as SABP block, which is a block placed at the height of the fifth intercostal in the medial/posterior axillary line between the anterior pterygoid muscle and the dorsal widest muscle.

In some cases, this allowed the procedure to be carried out due to patient burdens, relative contraindications and high risk of complications during general anesthesia. After studies related to the volume of local anesthetics administered as well as the concentration of their mixture, the optimal concentration of the substance used for regional blockade was chosen. This is a mixture of 0.125% ropivacaine solution with 0.25% lidocaine solution in a total volume of 60mL of administered solution.

Superficial parastenal intercostal plane block (SPIP) formerly known as TTP/ PIP/ PIFP/ SIP/ PSP which is an alternative combination in combination with SSAP is a block in which we deposit a local anesthetic in the parasternal line at the level of the 4th and 5th intercostal spaces between the internal intercostal muscle and the transverse thoracic muscle.

The purpose of the study is to determine whether SPIP+SSAP blockade is the optimal form of anesthesia for S-ICD implantation.

The patient, after qualifying by the cardiologist for S-ICD implantation, will undergo a standard anesthesiological qualification process with evaluation of basic demographic parameters, examination of body mass composition by bioimpedance, comorbidities, medications taken, determination of surgical risk according to the ASA scale ( American Society of Anesthesiology) in addition, the patient will be checked for any contraindications to the use of regional blockade as a method of anesthesia. After qualification, the patient will be asked to read the consent to participate in the study and sign the informed consent form.

Patients will receive standard premedication in the form of 1g of paracetamol and 150mg of pregabalin orally 30min before the procedure.

The subjects will be randomly divided into 2 groups - Group I will be patients administered PSP+SSAP anesthesia (consecutively 20+40ml of the mixture indicated above). Group II will be patients given SPIP+SSAP blockade ( consecutively 20+40ml of the mixture indicated above). It was tentatively planned to conduct the study on a group of 32 patients (16 in each of the two groups).

Anesthesiologists administering anesthesia prior to surgery receive an envelope with a randomly indicated method of anesthesia based on simple randomization determines the type of regional blockade used during the procedure). The subject will not know which study group he or she has been classified into. The operator performing the procedure will not be informed of the type of anesthesia performed -[randomization by double-blinding]. The operator performing the procedure will not be informed about the type of block performed in order to objectivize the extent and quality of the subject's anesthesia, which he will evaluate after the procedure according to a scale of subjective operator comfort created (EOA scale).

During the procedure, i.v. analgesia with the short-acting opioid remifentanil in the dose range of 0.025ug/kg/min to 0.1ug/kg/min will be administered as needed to control pain.

Increasing the dosage of the drug above these doses for pain control will be a disqualifying factor for the patient from further examination and the blockade will be considered ineffective which will be associated with receiving the lowest possible value on the operator's comfort scale. The use of i.v analgesics in the form of ketoprofen 100mg, metamizole 2.5g will also be allowed during the procedure.

During the procedure, the operator will be allowed to additionally administer local anesthesia to the area of the surgical field where severe pain is experienced. Infiltration of the surgical field with a solution of 1% lidocaine with epinephrine in a volume of no more than 40ml will then be performed If it is necessary to exceed the volume of local anesthesia, the patient will be disqualified from further examination. After the procedure, for the purpose of test defibrillation (checking the function of the implanted device), the patient will be put under short-term deeper sedation with propofol at a single dose of 1-3mg/kg/m.c. on one occasion.

During the procedure, in order to assess the patient's pain, NRS(numerical pain scale) or VAS(visual analog scale) scales will be checked every 15min. At the same intervals, the patient's level of sedation will be assessed using the RASS (Richmond agitation/sedation scale) and GCS (Glasgow level of consciousness) scales. Parameters such as SpO2 (hemoglobin oxygen saturation) NIBP( non-invasive blood pressure measurement) or HR (heart rate) will be monitored every 5min.

The NRS check in post-operative care will be done every 6h on the first day, the QoR-15 form (post-operative quality of life and improvement scale) will be given to the patient to fill in 24h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-90 years requiring S-ICD implantation for cardiac indications,
* high risk of anesthesia (ASA II or higher), patients giving informed consent to participate in the study.

Exclusion Criteria:

* absolute contraindications to regional anesthesia such as generalized coagulation disorders, inflammation at the site of anesthesia, allergy to the drugs used for regional anesthesia
* lack of consent of the patient for the conducted procedure,
* inability to cooperate with the patient - such as severe mental retardation, unregulated mental illness with motor agitation, advanced neurodegenerative diseases such as Parkinson's disease/Alzheimer's,
* inability to give informed consent to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
NRS | Checked at regular 15-minute intervals during the procedure and every 6 hours for the first 24 hours after the procedure
  numerical pain scale 0-10 points
VAS | Checked at regular 15-minute intervals during the procedure and every 6 hours for the first 24 hours after the procedure
  visual analogue scale 0-10 points
QoR - 15 | Administered to the patient before surgery and 24 hours after surgery
  post-operative quality of life and improvement scale 0-150 points
RASS | Checked at regular 15 minute intervals during the procedure
  Richmond arousal/sedation scale) (-5 <->+5) points
GCS | Checked at regular 15 minute intervals during the procedure
  Glasgow level of consciousness score scales 3-15 points
EOA | Checked immediately after the procedure (last suture)
  Effectiveness of Anaesthesia) -scale (-3 do +3) points

SECONDARY OUTCOMES:
SpO2 | Monitored every 5 minutes during the procedure
  hemoglobin oxygen saturation 50-99%
NIBP | Monitored every 5 minutes during the procedure
  non-invasive blood pressure measurement of 0-200 millimeters of the mercury column (mmHg)
HR | Monitored every 5 minutes during the procedure
  heart rate

OTHER OUTCOMES:
BMI | Before performing procedure
  Body mass index 15-45
bioimpedance | beforeperforming procedure
  volume od lipids 30-80%

CONTACTS AND LOCATIONS:
Overall Officials: Marek Szamborski, MD, Principal Investigator — Senior Assistant
Locations (1):
- 4th Military Clinical Hospital with Polyclinic, Wroclaw, Lower Silesian Voivodeship, Poland